CLINICAL TRIAL: NCT02285036
Title: A Phase III Clinical Trial for a Newly 23-valent Pneumococcal Polysaccharide Vaccine in Chinese Adults and Children
Brief Title: Safety and Immunogenicity of a Newly 23-valent Pneumococcal Polysaccharide Vaccine in Chinese Adults and Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Walvax Biotechnology Co., Ltd. (Industry)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government); Air Force Military Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Walvax-01
Record Dates: First submitted 2014-10-28; First posted 2014-11-06 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Pneumococcal Infectious Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A newly PPV23 (Experimental): The treatment pneumococcal vaccine was developed by Yunnan Walvax Biotech Co., Ltd (Walvax) China, is a sterile, liquid vaccine for intramuscular or subcutaneous injection. It consists of a mixture of highly purified capsular polysaccharides from the 23 most prevalent or invasive pneumococcal types of Streptococcus pneumoniae, including the six serotypes that most frequently cause invasive drug-resistant pneumococcal infections among children and adults in China. The dose of vaccine is an individual with a 0.5ml dose contains 23 kinds of pneumococcal polysaccharide serotypes each 25μg, and does not contain any preservatives. Vaccination of single dose of either treatment vaccine or control vaccine intramuscularly was performed in a ratio of 1:1.
  Interventions: Biological: vaccination PPV23
- PNEUMOVAX 23 (Active Comparator): PNEUMOVAX 23 is an established US-licensed vaccine and manufactured by the Merck Research Laboratories. Each 0.5 mL dose of vaccine contains 25μg of each polysaccharide type in isotonic saline solution containing 0.25% phenol as a preservative.Vaccination of single dose of either treatment vaccine or control vaccine intramuscularly was performed in a ratio of 1:1.
  Interventions: Biological: vaccination PNEUMOVAX 23

INTERVENTIONS:
Biological: vaccination PPV23 — All eligible participants were stratified into four age strata namely, 2 to 6 years, 7 to 17 years, 18 to 59 years and more than 60 years. Stratified, block randomization with a size of eight was applied. Vaccination of single dose of either treatment vaccine or control vaccine intramuscularly was performed in a ratio of 1:1. Blood samples were obtained from each subject at baseline, day 30-35 after injection, to evaluate immunogenicity.
  Arms: A newly PPV23
Biological: vaccination PNEUMOVAX 23 — Vaccination of single dose of either treatment vaccine or control vaccine intramuscularly was performed in a ratio of 1:1.
  Arms: PNEUMOVAX 23

SUMMARY:
A newly 23-valent pneumococcal polysaccharide vaccine was developed with promising safety and immunogenicity demonstrated in the phase III trial in China. A large scale, double blind, randomized, PNEUMOVAX 23 (Merck & Co., Inc.) controlled phase 3 clinical trial was conducted.

DETAILED DESCRIPTION:
The World Health Organization (WHO) estimated that more than 800 000 children younger than 5 years died from pneumococcal disease in 2000, making it the leading vaccine-preventable cause of death. Pneumococcal polysaccharide vaccines have progressed from 2-valent vaccines to the current 23-valent vaccine, which has been available since the early 1980s. The 23-valent vaccine includes serotypes accounting for 72% to 95% of invasive pneumococcal disease, depending on the geographic area. Many countries have added pneumococcal polysaccharide vaccine to their existing national immunization programs or recommended it for people aged 65 years and older and for individuals aged 2-64 who are at increased risk of pneumococcal disease.

A newly 23-valent pneumococcal polysaccharide vaccine was developed with promising safety and immunogenicity demonstrated in the phase III trial in China. A large scale, double blind, randomized, PNEUMOVAX 23 (Merck & Co., Inc.) controlled phase 3 clinical trial was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants older than 2 years were recruited and enrolled in September or October 2012.
* Participants with axillary temperature less than Celsius 37 degrees
* Not yet having received pneumococcal vaccine and other prevention products within 7 days.

Exclusion Criteria:

* Exclusion criteria were any known primary or secondary immunodeficiency
* Allergy
* Severe cardiovascular disease bleeding disorders
* Receipt of immunoglobulin or blood products within one month and so on.-

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1660 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
the rate of 2-fold increase of anti-pneumococcal antibody | 30 days after the injection of vaccination

SECONDARY OUTCOMES:
geometric mean concentration (GMC) | 30 days after the injection of vaccination
geometric mean fold increase (GMFI) | 30 days after the injection of vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Yanping Li, Principal Investigator — Guangxi Provincial Center for Diseases Control and Prevention
Locations (1):
- Guangxi Provincial Center for Diseases Control and Prevention, Nanning, Guangxi, China